CLINICAL TRIAL: NCT00562614
Title: A Pilot Phase IIa Randomised, Double-blind, Placebo-controlled, Crossover Study to Examine the Safety, Tolerability and Pharmacodynamic Effects on Blood Pressure of Repeat Oral Doses of SLx-2101 5 mg or 10 mg Once Daily for up to 14 Days in Patients With Hypertension
Brief Title: Safety and Effect of Oral Doses of 5mg or 10mg of SLx-2101 for 14 Days in Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-2101-07-08
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2015-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLx-2101
  Interventions: Drug: SLx-2101
- 2 (Placebo Comparator): Comparative Placebo Dose
  Interventions: Drug: SLx-2101

INTERVENTIONS:
Drug: SLx-2101

SUMMARY:
The purpose is to determine the effect of SLx-2101 dosed at 5mg or 10mg for 14 days on systolic, diastolic pressures and heart rate in patients with hypertension.

DETAILED DESCRIPTION:
1. Placebo-corrected supine peripheral systolic, diastolic blood pressures and heart rate
2. 24 hour ambulatory blood pressure and heart rate
3. Safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 70 years old, inclusive
* Moderate to severe hypertension
* Body weight within a body mass index of 18-32kg/m2

Exclusion Criteria:

* The subject is receiving more than three antihypertensive agents
* A history of drug abuse
* Exposure to a new chemical entity within 3 months prior to the first day of dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Peripheral systolic, diastolic blood pressures and heart rates | 14 days

SECONDARY OUTCOMES:
Adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, MD, Principal Investigator — PAREXEL, Institute for Clinical Pharmacology
Locations (1):
- Parexel, Institute for Clinical Pharmacology, Berlin, Germany